CLINICAL TRIAL: NCT00287560
Title: A Comparison of Venous Tolerability and Injection Pain of a Modified Propofol Preparation and Standard Propofol in the Induction of Anesthesia in Children
Brief Title: Effect of a Modified Propofol Preparation on Injection Pain During Induction of Anesthesia in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: B. Braun Melsungen AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BBMDE-0312
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2008-02-25 (Estimated); Status verified 2008-02

CONDITIONS: Anesthesia
MeSH Terms: interventions — Propofol; Pharmaceutical Preparations

INTERVENTIONS:
Drug: propofol (drug)

SUMMARY:
The purpose of the study is to determine wether a modified propofol preparation shows any effect on the incidence of injection pain in children undergoing elective surgery under general anesthesia.

Study hypothesis: The use of a modified propofol preparation will reduce the incidence of injection pain in the study group.

DETAILED DESCRIPTION:
Pain on injection is the most frequently reported side effect associated with the use of propofol for induction of anesthesia. Various measures have been taken to reduce the pain on injection, e.g. administration of lidocaine or fentanyl prior to propofol administration, mixture of lidocaine and propofol as well as cooling of the emulsion. Although pain on injection had been reduced with some of the above mentioned methods, they may not be regarded as a satisfactory solution of the problem.

ELIGIBILITY:
Inclusion Criteria:

* age >= 2 and < 6 years
* written informed consent of the parents
* anesthetic risc classified as ASA I - III
* patient undergoing elective surgery under general anesthesia
* venous access for induction of anesthesia on the dorsum of the hand
* hospital care for at least 3 hrs after end of anesthesia guaranteed

Exclusion Criteria:

* intolerability of the drugs tested
* current drug medication with sedative effect
* patient is expected to require concomitant medication not allowed in the study
* history of or current renal or hepatic disease, cardiac insufficiency
* hypovolemia
* increased cranial pressure
* simultaneous participation in another clinical trial or participation during the month preceding this study

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64
Dates: Start 2003-08; Study Completion 2005-02

PRIMARY OUTCOMES:
incidence of spontaneous expression of pain during injection

SECONDARY OUTCOMES:
anesthetists VAS for assessment of injection pain, propofol dosage and requirements, hemodynamic parameters, safety laboratory, adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Gerd P Molter, MD, PhD, Principal Investigator — Klinik für Anästhesie und operative Intensivmedizin, Klinikum Leverkusen gGmbH